CLINICAL TRIAL: NCT06212908
Title: Integrating Periodontal Therapy and Biofilm Management Into Breast Cancer Patients' Care: Periodontal, Hematological and Salivary Parameters Assessment Before and During Chemotherapy
Brief Title: Assessment of Periodontal Therapy and Biofilm Management in Breast Cancer
Acronym: BREASTCANCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Daniela Bazan Palioto (Unknown)
Responsible Party: Principal Investigator, Kelly Rocio Vargas Villafuerte, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 03121212.6.3001.5440
Record Dates: First submitted 2023-12-30; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Gingivitis; Periodontal
Keywords: Breast cancer; Gingivitis; Periodontal therapy
MeSH Terms: conditions — Breast Neoplasms; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer (Other): The division was made into 2 groups: Patients with breast cancer and gingivitis (BC/G) (n=20); and control patients with gingivitis only (G) (n=20).
  Clinical periodontal examinations were carried out by a single trained and calibrated examiner. Clinical periodontal, hematological and salivary flow parameters were assessed at baseline, 6 weeks, 12 and 24 weeks.
  Interventions: Other: Basic Periodontal Therapy

INTERVENTIONS:
Other: Basic Periodontal Therapy — All patients received oral hygiene instructions (interproximal cleaning with floss and interdental brushes, brushing instructions on the Bass technique). The patients were also encouraged to brush the back of the tongue once a day. Subsequently, all patients underwent supragingival scaling, prophylaxis, and polishing. Supragingival scaling was performed using manual instruments (Gracey curettes) and an ultrasonic device.
  Other Names: Biofilm control

SUMMARY:
Objective: To evaluate the impact of chemotherapy on periodontal conditions, hematology, and salivary flow in patients with breast cancer and gingivitis, after basic periodontal therapy (BPT).

Methods: They were divided into patients with breast cancer and gingivitis (BC/G =20); and patients without cancer with gingivitis (G=20). Clinical parameters [Plaque Index (PI), bleeding on probing (BOP), Probing Depth (PS), Clinical Attachment Level (CAL)], hematological parameters (complete blood count), and salivary flow were evaluated at baseline, 6, 12 and 24 weeks.

DETAILED DESCRIPTION:
Objective: To evaluate the impact of chemotherapy on periodontal conditions, hematology, and salivary flow in patients with breast cancer and gingivitis, after basic periodontal therapy (BPT).

Methods: They were divided into patients with breast cancer and gingivitis (BC/G =20); and patients without cancer with gingivitis (G=20). Clinical parameters [Plaque Index (PI), bleeding on probing (BOP), Probing Depth (PS), Clinical Attachment Level (CAL)], hematological parameters (complete blood count), and salivary flow were evaluated at baseline, 6, 12 and 24 weeks.

ELIGIBILITY:
- All patients were diagnosed with localized gingivitis (G) The inclusion criteria were: At least 15 teeth; no loss of attachment and probing depth ≤ 3mm; bleeding on probing ≥ 10% of sites, no radiographic bone loss.

Exclusion Criteria:

1) systemic diseases (e.g. diabetes, cardiovascular diseases) or autoimmune diseases in addition to cancer; 2) patients with periodontitis; 3) use of any medication that could interfere with periodontal aspects; 4) smokers; 5) Pregnant or lactating patients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer
Enrollment: 40 (Actual)
Dates: Start 2012-09-18 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Periodontal conditions | before and after post treatment (baseline, 6 weeks, 12 and 24 weeks)
  The plaque index (PI) was determined by analyzing the presence or absence of biofilm on the gingival margin, expressed as a percentage of surfaces with biofilm Bleeding on probing (BOP) was determined by detecting the presence or absence of bleeding, expressed as the percentage of bleeding surfaces.
  The probing depth (PD/mm) was expressed in millimeters, measured from the gingival margin to the bottom of the gingival sulcus.
  The clinical attachment level (CAL/mm) was expressed in millimeters, measured from the cementoenamel junction to the most apical portion of the gingival sulcus.
  Both BOP, PD, CAL were evaluated at six locations per tooth, i.e., three on the buccal surface and three on the lingual or palatal surface.
  Periodontal parameters (BOP, PD, CAL and PI ) are evaluated together or combined to perform periodontal diagnosis

SECONDARY OUTCOMES:
Salivary Flow | before and after post treatment (baseline, 6 weeks, 12 and 24 weeks)
  The salivary flow rate was expressed in milliliters per minute (mL/min). Periodontal parameters and salivary flow will be combined to assess oral health.